CLINICAL TRIAL: NCT03784339
Title: Feasibility Study: Does a Designated Education Session Change Levels of Catastrophizing, Kinesiophobia and Pain Beliefs in Patients With Patellofemoral Pain?
Brief Title: Effect of Designated Education Session on Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, James Selfe, DSc, Professor of Health Professions, Manchester Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PatellofemoralPain_DEC2018
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Knee Cap
Keywords: Patellofemoral; Knee
MeSH Terms: conditions — Patella Fracture | interventions — Physical Therapy Modalities; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy (Placebo Comparator): Participants will receive standard physiotherapy care, which will involve strength exercises and taping.
  Interventions: Other: Physiotherapy
- Physiotherapy + education (Experimental): Physiotherapy + education Standard physiotherapy care plus 30 minute education session addressing fear of movement and catastrophizing thoughts.
  Interventions: Other: Physiotherapy + education; Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy + education — Participants will take part in a 30 minute education session surrounding fear of movement and catastrophizing thoughts. They will then receive standard care, which will involve strength exercises and taping if needed.
  Arms: Physiotherapy + education
Other: Physiotherapy — Standard physiotherapy care

SUMMARY:
Feasibility study: Does a designated education session change levels of catastrophizing, kinesiophobia and pain beliefs in patients with patellofemoral pain? Design: Single site feasibility Study Aim: Aims are to identify if a formal education session (intervention) improves patient outcomes and to assess if it is possible to test the intervention for efficacy in a larger study.

Outcome Measures: The primary outcome measure is the Knee Osteoarthritis Outcome Score-Patellofemoral) KOOS-PF. The original KOOS consists of 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of Life (QOL). The KOOS-PF was developed to evaluate individuals or samples of individuals who present with anterior knee pain/patellofemoral pain and/or patellofemoral osteoarthritis (OA), or who are at risk of developing patellofemoral pain or OA.

Secondary Outcome Measures are Pain Catastrophizing Scale and The Tampa Scale for Kinesiophobia.

Patients who are eligible for inclusion in the study will be identified from the Musculoskeletal Clinical Assessment Service (MCAS) by Band 6's and 7's and approved by a Band 8 Physiotherapist the South Liverpool Treatment Centre.

Intervention: The intervention will comprise a 1:1, 30 minute education session delivered by a specialist musculoskeletal physiotherapist with over ten years' experience who has an interest in patellofemoral pain.

The education session will be based on a schedule formed from the most recent research on patellofemoral pain PFP which considers psychosocial factors (Robertson et al 2017). Crepitus is a word used to describe any grinding, creaking, cracking, grating, crunching or popping that occurs when the patellofemoral joint moves (Robertson et al 2017). The psychological factors, specifically patients' beliefs about crepitus, avoiding crepitus and the influence of others will be discussed.

The intervention will be supported by the leaflet 'managing my patellofemoral pain' developed by Barton and Rathleff (2016) on the basis of international opinion from 21 international experts and subsequent review by 20 patients diagnosed with PFP to ensure clarity.

Duration: Within the time constraints of a Masters Degree, patients will be recruited over a four month period. There will be four months for follow up and a further four months for write up, total study duration 12 months.

DETAILED DESCRIPTION:
Design: A feasibility study to assess if a physiotherapy education session in addition to standard care improves patients scores regarding catastrophizing and kinesiophobia when measured by KOOS-PF, Pain Catastrophizing Scale and Tampa Scale

Objectives:

1. To assess if providing a specific education session which reviews patients beliefs about crepitus, causes of pain, joint mechanics and purpose of exercise has an effect on catastrophizing and kinesiophobia.
2. To identify if the study is feasible on a larger scale, which would allow the intervention to be assessed for efficacy. If a future study was able to demonstrate that the intervention was effective this would provide an additional evidence based intervention for use in clinical practice.

Recruitment: NHS patients diagnosed in a Musculoskeletal Clinical Assessment Service [MCAS] with patellofemoral pain at the South Liverpool Treatment Centre.

Inclusion criteria:

* Adults aged 18-40
* Be able to understand and converse in English
* Clinical diagnosis of PFP
* Be able to attend for up-to 12 weeks of physiotherapy

Exclusion criteria:

* Patients who present with referred pain from the spine or hip, or have tibiofemoral pathology of any nature on the ipsilateral side.
* A diagnosis of patellofemoral joint (PFJ) OA as confirmed by X-Ray or Magnetic Resonance Imaging (MRI).

Sample size: There is limited published research regarding the use of the questionnaire KOOS-PF in research. As a result it is not possible to do a definitive study to test whether or not the education session effects patient outcome. Therefore it is necessary to do a feasibility study with a small sample size of 24 patients (control n=12, intervention n=12) which will allow any change in the questionnaire scores to be used to calculate how many patients would be needed for a definitive study which would allow researchers to assess whether or not the exercise intervention affected patient outcome, which could improve patient care. The research team are confident that the required number of patients could be recruited as audit data from the service identified that 104 patients in the MCAS service met the criteria for inclusion in this proposed study.

Baseline measures: Participants' characteristics including age, gender and duration of symptoms will be collected alongside baseline measures for the chosen questionnaires - the KOOS-PF, Tampa-scale for Kinesiophobia and Pain Catastrophizing. These questionnaires will be repeated at 12 weeks.

Intervention: Patients recruited into the study will be randomised to either the intervention (n=12) or the control group (n=12). Participants in the control group will undergo standard treatment.

The intervention: Participants in the intervention group will receive standard treatment plus the education session.

The education session will be based on a leaflet produced by other leading researchers in the field and will also explore the causes of pain, beliefs about pain, beliefs about noise that come from the joint, the impact of the pain on activity and the influence of other family members' experience and beliefs about knee pain. At 12 weeks, participants from both groups will be asked to repeat the questionnaires.

Statistical analysis: Descriptive statistical analysis will be performed on the data and the lead researcher will work with the statistics department at MMU to review the change in the chosen questionnaires to identify the sample size required for a definitive study which will assess how effective the education session is on patients' symptoms of PFP.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-40
* Be able to understand and converse in English
* Clinical diagnosis of PFPS
* Be able to attend for up-to 12 weeks of physiotherapy

Exclusion Criteria:

* Patients who present with referred pain from the spine or hip, or have tibiofemoral pathology of any nature on the ipsilateral side.
* A diagnosis of PFJ osteoarthritis as confirmed by X-Ray or MRI.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Knee Osteoarthritis Outcome Score - Patellofemoral (KOOS-PF) | 12 weeks following baseline visit
  The KOOS-PF is an 11 item, patient reported outcome measure of pain and function where a maximum score of 100 indicates no problems and a minimum score of 0 indicates extreme problems.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK) | 12 weeks following baseline visit
  The TSK is a 17-item patient reported outcome measure of fear of movement. A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible. A score of 68 is the highest possible score and indicates extreme fear of pain with movement.
Pain Catastrophizing Scale (PCS) | 12 weeks following baseline visit
  The PCS is a 13 item patient reported outcome measure where the PCS total score is computed by summing the responses to all 13 items. PCS total scores range from 0 - 52, with higher scores indicating greater pain catastrophizing

CONTACTS AND LOCATIONS:
Overall Officials: James Selfe, Study Chair — Professor
Locations (1):
- Royal Liverpool & Broadgreen University Hospitals Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No